CLINICAL TRIAL: NCT04329000
Title: The Impacts of On-demand Versus Continuous Esomeprazole Therapy on the Symptom Control and Histological Changes of Metaplastic Esophageal Epithelium in Patients With Barrett's Esophagus (EsoBE) - a Multicentre Randomized Controlled Trial
Brief Title: On-demand PPI Therapy is Effective on Controlling Symptoms in Patients With Barrett's Esophagus.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Sung-shuo Kao, Principal Investigator, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VGHKSBE01
Record Dates: First submitted 2020-03-25; First posted 2020-04-01 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Barrett Esophagus; Proton Pump Inhibitor; Symptom; Reflux
Keywords: Barrett's Esophagus; Erosive esophagitis; Proton pump inhibitor; On-demand therapy; Continuous therapy
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Intervention Model Description: Randomized-controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- On-demand PPI therapy (Experimental): The patients in this group were advised to take PPI for 8 weeks continuously, followed by on-demand PPI therapy for the following 40 weeks.
  Interventions: Drug: Esomeprazole 40mg
- Continuous PPI therapy (Active Comparator): The patients in this group were advised to take PPI QD continuously for 48 weeks.
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole 40mg — On-demand Esomeprazole 40 mg QD
  Other Names: nexium 40 mg
  Arms: On-demand PPI therapy
Drug: Esomeprazole — Continuous Esomeprazole 40 mg QD
  Other Names: nexium 40 mg
  Arms: Continuous PPI therapy

SUMMARY:
On-demand PPI therapy is feasible for the long-term treatment of patients with Barrett's esophagus.

DETAILED DESCRIPTION:
Consecutive patients with symptomatic Barrett's esophagus are recruited and receive biopsy for esophageal metaplastic mucosa and gastric mucosa over the antrum and body during endoscopy on enrollment. The biopsy protocol for esophageal metaplastic mucosa is following Seattle protocol. GERD Q score will be conducted on enrollment. Additionally, blood sampling for CYP2C19 genotyping is also conducted on enrollment. The eligible subjects will be treated by 8-week esomeprazole, and are then randomly assigned to receive either maintenance or on-demand esomeprazole therapy (40 mg q.d.) for 40 weeks. The patients were asked to come back every four weeks for the recording of symptom days and PPI tablet consumption numbers. Follow-up endoscopy with biopsy for esophageal and gastric mucosa is performed at the end of the 48th weeks. We will compare the effects of maintenance and on-demand PPI therapy on (1) histological changes of esophageal metaplastic mucosa (2) symptom control (3) tablet consumption number

ELIGIBILITY:
Inclusion Criteria:

* patients between the ages of 20 and 80 years
* having symptoms of acid regurgitation, heart burn, or feeling of acidity in the stomach
* having Barrett's Esophagus proven by histology confirmation
* length of esophageal metaplastic mucosa equal to or longer than 1 centimeter

Exclusion Criteria:

* pregnancy,
* coexistence of serious concomitant illness (for example, decompensated liver cirrhosis and uremia)
* previous gastric surgery,
* allergic to esomeprazole,
* presence of dysplastic esophageal mucosa
* equivocal endoscopic diagnosis of Barrett's esophagus

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 218 (Actual)
Dates: Start 2010-02-02 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-12-08 (Actual)

PRIMARY OUTCOMES:
Rates of progression, remaining unchanged, or regression of the distal esophageal metaplastic mucosa in both groups after 48 weeks | 48 weeks.
  Progression, stationary, regression
Total symptom day | 48 weeks
  Days with reflux symptoms
Number of tablets consumed | 48 weeks
  PPI tablets consumed during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: SUNG-SHUO KAO, Bachelor, Principal Investigator — Kaohsiung Veterans General Hospital.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kahrilas PJ. Clinical practice. Gastroesophageal reflux disease. N Engl J Med. 2008 Oct 16;359(16):1700-7. doi: 10.1056/NEJMcp0804684. PMID 18923172
- [Background] Vakil N, van Zanten SV, Kahrilas P, Dent J, Jones R; Global Consensus Group. The Montreal definition and classification of gastroesophageal reflux disease: a global evidence-based consensus. Am J Gastroenterol. 2006 Aug;101(8):1900-20; quiz 1943. doi: 10.1111/j.1572-0241.2006.00630.x. PMID 16928254
- [Background] Attwood SE, Lundell L, Hatlebakk JG, Eklund S, Junghard O, Galmiche JP, Ell C, Fiocca R, Lind T. Medical or surgical management of GERD patients with Barrett's esophagus: the LOTUS trial 3-year experience. J Gastrointest Surg. 2008 Oct;12(10):1646-54; discussion 1654-5. doi: 10.1007/s11605-008-0645-1. Epub 2008 Aug 16. PMID 18709511
- [Background] Kastelein F, Spaander MC, Steyerberg EW, Biermann K, Valkhoff VE, Kuipers EJ, Bruno MJ; ProBar Study Group. Proton pump inhibitors reduce the risk of neoplastic progression in patients with Barrett's esophagus. Clin Gastroenterol Hepatol. 2013 Apr;11(4):382-8. doi: 10.1016/j.cgh.2012.11.014. Epub 2012 Nov 28. PMID 23200977
- [Background] Laine L, Ahnen D, McClain C, Solcia E, Walsh JH. Review article: potential gastrointestinal effects of long-term acid suppression with proton pump inhibitors. Aliment Pharmacol Ther. 2000 Jun;14(6):651-68. doi: 10.1046/j.1365-2036.2000.00768.x. PMID 10848649
- [Background] Sharma P, Dent J, Armstrong D, Bergman JJ, Gossner L, Hoshihara Y, Jankowski JA, Junghard O, Lundell L, Tytgat GN, Vieth M. The development and validation of an endoscopic grading system for Barrett's esophagus: the Prague C & M criteria. Gastroenterology. 2006 Nov;131(5):1392-9. doi: 10.1053/j.gastro.2006.08.032. Epub 2006 Aug 16. PMID 17101315
- [Background] Gatenby PA, Ramus JR, Caygill CP, Shepherd NA, Watson A. Relevance of the detection of intestinal metaplasia in non-dysplastic columnar-lined oesophagus. Scand J Gastroenterol. 2008;43(5):524-30. doi: 10.1080/00365520701879831. PMID 18415743

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT04329000/Prot_SAP_000.pdf